CLINICAL TRIAL: NCT06475053
Title: Visual Performance of Center Distance Daily Disposable Multifocal Lenses
Acronym: ViPCD3
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Visioneering Technologies, Inc (Industry)
Collaborators: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: VTI-2405
Record Dates: First submitted 2024-06-04; First posted 2024-06-26 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Myopia
Keywords: Contact lens; Multifocal
MeSH Terms: conditions — Myopia | interventions — Contact Lenses

STUDY DESIGN:
Intervention Model Description: This will be a prospective, double-masked, crossover trial.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and the examiner tasked with obtaining study outcome data will be masked to the design or brand of lenses. An unmasked examiner will be available to address any issues of lens wear or other adverse events.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- NaturalVue (Active Comparator): NaturalVue Enhanced Multifocal 1 Day contact lens
  Interventions: Device: NaturalVue Enhanced Multifocal 1 Day contact lens
- MiSight (Active Comparator): MiSight 1 Day contact lens
  Interventions: Device: MiSight 1 Day contact lens

INTERVENTIONS:
Device: NaturalVue Enhanced Multifocal 1 Day contact lens — Daily disposable multifocal contact lens
  Arms: NaturalVue
Device: MiSight 1 Day contact lens — Daily disposable dual-focus contact lens
  Arms: MiSight

SUMMARY:
The purpose of this study is to compare visual performance (high and low contrast acuity, reading acuity, contrast sensitivity, stereoacuity, accommodative response, eye hand coordination, far near vision, and dynamic vision) between Visioneering Technologies, Inc. NaturalVue Multifocal and CooperVivion MiSight.

ELIGIBILITY:
Inclusion Criteria:

* Participants must satisfy the following conditions for inclusion in the trial:

  * Be between 9 and 30 years of age
  * Sign written Informed Consent/Assent.
  * Spherical Equivalent glasses prescription: -0.50 to -7.00 diopters (D), Astigmatism: ≤ -0.75D, Anisometropia: ≤ 1.00D
  * 20/20 vision in each eye
  * Existing contact lens wearer
  * An eye exam in last 9 months, normal stereoacuity on prior chart (or test if not available)
  * No known ocular disease - anterior or posterior (posterior determined by history/chart)
  * Have an acceptable or optimal fit with test lenses and be willing to wear these lenses as directed for the duration of the study.
  * On examination, have ocular findings considered to be within normal limits.
  * Be willing and able to follow instructions and attend the schedule of follow-up visits.

Exclusion Criteria:

* Any of the following will exclude a participant from this trial:

  * Current hard lens wearers
  * Using eye medication contraindicating lens wear such as daily use of artificial tears.
  * Eye injury or surgery within twelve weeks immediately prior to enrollment for this trial.
  * History of corneal refractive surgery
  * Currently enrolled in an ophthalmic clinical trial that could negatively impact corneal or conjunctival health in this trial.
  * Evidence of systemic or ocular abnormality, infection or disease likely to affect successful wear of contact lenses or use of their accessory solutions.
  * Allergy or sensitivity to any product used in this trial.
  * Pre-existing ocular condition that would contraindicate lens wear.
  * Any systemic disease including autoimmune disease, immunocompromising diseases, connective tissue disease, clinically significant atopic diseases, insulin dependent diabetes, use of medications including corticosteroids and antimetabolites that may affect the eye or be exaggerated by wearing contact lenses.
  * Lazy eye (Strabismus or amblyopia)
  * Pupil size < 3.00 mm in either eye in dim light (measured at approximately 10 cd/m2 )

Ages: 9 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of visual performance (high and low contrast acuity) between VTI NaturalVue Enhanced Multifocal and CooperVision MiSight. | 2 months
  log MAR vision scale

CONTACTS AND LOCATIONS:
Overall Officials: Marjean T Kulp, OD, MS, Principal Investigator — The Ohio State University College of Optometry
Locations (1):
- The Ohio State University College of Optometry, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No